CLINICAL TRIAL: NCT02707744
Title: A Prospective Observational Study of Prolonged Electrocardiographic Monitoring in Patients With Heart Failure in Sinus Rhythm or Atrial Fibrillation
Brief Title: A Study of Prolonged Electrocardiographic Monitoring in Patients With Heart Failure in Sinus Rhythm or Atrial Fibrillation
Acronym: POP-ECG-HF-AF
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15IC2955
Record Dates: First submitted 2016-02-08; First posted 2016-03-14 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: Heart Failure; Atrial Fibrillation; Ambulatory ECG monitor
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sinus rhythm: patients with heart failure and sinus rhythm
  Interventions: Other: no intervention
- atrial fibrillation: patients with heart failure and atrial fibrillation
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
It is an observational study in patients with heart failure investigating the incidence of arrhythmias using a wearable device which can monitor heart rhythm for up to 14 days. In addition to gathering routine clinical information, research assessments include a symptoms questionnaire and a corridor walk test. Patients will be followed for clinical events (interventions for arrhythmias, hospitalisation, death) for 1 year.

DETAILED DESCRIPTION:
due to the slow recruitment, on the one hand, and the fact that the preliminary analysis gave the valuable results, on the other hand, the number of patients was reduced from 400 to 100 and the follow-up from five years to one year

ELIGIBILITY:
Inclusion Criteria:

1. Heart Failure
2. Treated with Loop Diuretics for at least six weeks
3. Willing and legally able to sign informed consent
4. At least 18 years of age
5. New York Heart Association (NYHA) class II - IV

Exclusion Criteria:

1. Myocardial infarction in the previous six weeks,
2. Implanted pacemaker, including cardiac resynchronisation device, or defibrillator
3. Already participating in an interventional randomized controlled trial assessing effects on morbidity and mortality (this study does not preclude participation in future clinical trials).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with heart failure
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Greater Glasgow and Clyde, Glasgow
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Northwick Park Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sinus Rhythm: patients with heart failure and sinus rhythm
  no intervention
- Atrial Fibrillation: patients with heart failure and atrial fibrillation
  no intervention
Period: Overall Study
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Started | 50 | 50
Completed | 47 | 50
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sinus Rhythm | Atrial Fibrillation | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [60 to 78] | 78 [74 to 83] | 75 [66 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 35 | 33 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 38 | 48 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 47 | 50 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Identified Dysrhythmia on Baseline ECG Recording
Description: A dysrhythmia will be defined as either
  1. Arrhythmia for which there is a Class I or IIa recommendation for treatment with medication or devices in ESC guidelines.
  2. One or more of the following even if it does not otherwise meet guideline-indication for treatment:
     * Sinus bradycardia ≤30bpm for ≥one minute
     * High-degree atrioventricular (AV) block (3rd degree or Mobitz Type I or II)
     * Pauses lasting ≥3 seconds (either sinus or AV block)
     * Frequent ventricular ectopy defined as >1,000 ectopic beats per day.
     * Ventricular tachycardia with rate ≥100 bpm for ≥5 beats.
Time Frame: on enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Number analyzed (Participants) | 47 | 50
Participants | 25 | 35

2. Secondary Outcome: Combined Endpoint Made up of Cardiovascular Mortality or Hospitalisation for the Management of Heart Failure/Arrhythmia or Implantation of Any Permanent Device Capable of Pacing the Heart.
Description: information about new implantations and hospitalisations were known for 46 patients with sinus rhythm (97.9%) and 47 with atrial fibrillation (94%)
Time Frame: From date of enrollment until the date of first hospitalization for management of heart failure/arrhythmia or date of implantation of any permanent device capable of pacing the heart or cardiovascular death, whichever came first, assessed up to 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Number analyzed (Participants) | 46 | 47
Participants | 24 | 18

3. Secondary Outcome: All Cause Mortality
Description: survival status was known in 46 patients with sinus rhythm (97.9%) and 50 patients with atrial fibrillation (100%)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Number analyzed (Participants) | 46 | 50
Participants | 3 | 4

4. Secondary Outcome: Cardiovascular Mortality
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Total Number of Hospitalisations for the Management of Heart Failure or Arrhythmia
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Total Number of Patients Implanted With Any Permanent Device Capable of Pacing the Heart
Description: information about new implantations were known for 46 patients with sinus rhythm (97.9%) and 47 with atrial fibrillation (94%)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Number analyzed (Participants) | 46 | 47
Participants | 16 | 7

7. Secondary Outcome: Implantation of Any Permanent Device Capable of Pacing the Heart
Description: as for outcome 6
Time Frame: From date of enrollment until the date of implantation of any permanent device capable of pacing the heart, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sinus Rhythm | Atrial Fibrillation
Number analyzed (Participants) | 46 | 47
Participants | 16 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sinus Rhythm | Atrial Fibrillation
All-Cause Mortality (participants affected / at risk) | 3/46 | 4/50
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 0/47 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02707744/Prot_SAP_ICF_000.pdf